CLINICAL TRIAL: NCT04169438
Title: "Randomized, Double-blind, Comparative Pilot Study Investigating the Safety and Clinical Efficacy of Applying a Restorative Wound Care Cream Together With Petrolatum on Anatomically Similar Surgical Excisions"
Brief Title: Pilot Study Investigating a Restorative Wound Care Cream Together With Petrolatum on Surgical Excisions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Center for Clinical and Cosmetic Research (Other)
Collaborators: BirchBioMed Inc. (Unknown)
Responsible Party: Principal Investigator, Mark Steven Nestor, M.D., Ph.D., Director, The Center for Clinical and Cosmetic Research
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: POC-1FLL
Record Dates: First submitted 2019-11-15; First posted 2019-11-19 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Wound Heal; Scar; Keloid; Surgical Wound
Keywords: Wound Heal; Scar; Keloid; Surgical Wound
MeSH Terms: conditions — Cicatrix; Keloid; Surgical Wound | interventions — Petrolatum

STUDY DESIGN:
Intervention Model Description: The study consists of two (2) Treatments, both of which are administered in combination with petrolatum. The Treatments consist of either a restorative wound care cream (FS2 ingredient) or a vehicle wound care cream (without the FS2 ingredient).
Who Masked: Participant, Investigator
Masking Description: This pilot study is double-blinded, which means that neither the evaluating physician nor the subject will know which treatment is administered. A separate study team member will administer the treatment as well as answer questions and discuss any problems throughout the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vehicle Cream Base Emulsion Moisturizer + Petrolatum (Placebo Comparator): Vehicle Cream Base Emulsion Moisturizer + Petrolatum
  Interventions: Other: Vehicle Cream Base Emulsion Moisturizer + Petrolatum
- FS2 Emulsion Moisturizer + Petrolatum (Experimental): FS2 Emulsion Moisturizer + Petrolatum
  Interventions: Other: FS2 Emulsion Moisturizer + Petrolatum

INTERVENTIONS:
Other: Vehicle Cream Base Emulsion Moisturizer + Petrolatum — Topical vehicle white (bone) color, oil/water emulsion moisturizer.
  Arms: Vehicle Cream Base Emulsion Moisturizer + Petrolatum
Other: FS2 Emulsion Moisturizer + Petrolatum — Topical FS2 white (bone) color, oil/water emulsion moisturizer.
  Arms: FS2 Emulsion Moisturizer + Petrolatum

SUMMARY:
The pilot study is prospective, randomized, double-blinded, with intra-subject comparisons against a vehicle control. The primary objective of this pilot study is to investigate the safety and effectiveness of a new wound care product formulated to improve healing outcome, minimize complications of impaired healing and minimize the appearance of scars.

This pilot study is double-blinded, which means that neither the evaluating physician nor the subject will know which treatment is administered.

Subjects' with 2 comparable excision sites will be randomly assigned to use the FS2 restorative wound care product on one excision site and a vehicle formulation of the product on the other. At the discretion of the Principal Investigator, a sutured wound may be bisected for intra-wound comparison of treatments. In all cases, after application of either vehicle or FS2, a layer of petrolatum will be applied to cover the wound site as a standard of care.

DETAILED DESCRIPTION:
The pilot study is prospective, randomized, double-blinded, with intra-subject comparisons against a vehicle control. The primary objective of this pilot study is to investigate the safety and effectiveness of a new wound care product formulated to improve healing outcome, minimize complications of impaired healing and minimize the appearance of scars. Per protocol, study team members will investigate the efficacy of applying investigational product in combination with petrolatum on similar anatomically matched surgical excisions and bisected sutured wounds for a period of up to 180 days.

Secondary to direct complications that arise from removal of a skin lesion is the aesthetic disfigurement of tissue repair that results in a scar. The severity of even the most morbid scars is unpredictable and largely dependent on several variables. It is for this reason that this pilot study seeks to evaluate the application of a wound care product on both sutured and un-sutured surgical wounds across all phases of wound healing.

General and widely commercialized self-care (OTC) wound healing products include emollients, lotions, petrolatum creams, and topical antibiotics. With only a limited number of investigator-initiated studies, the advancement in this niche medical sector has been incremental across decades of research. This study is being undertaken to investigate the safety and effectiveness of a new cream product (FS2-cream) which was initially intended to manage hyperproliferative closed scars by maintaining an optimal skin environment. To obtain proof-of-concept results that enable the robust design of subsequent studies, we will obtain wound care metrics across all phases of healing and make intra-subject comparisons between the use of FS2-cream + petrolatum and vehicle-cream + petrolatum. We hypothesize that FS2-cream + petrolatum will show superior clinical outcomes compared to the vehicle control treatment.

This pilot study is double-blinded, which means that neither the evaluating physician nor the subject will know which treatment is administered. A separate study team member will administer the treatment as well as answer questions and discuss any problems throughout the study.

Subjects' with 2 comparable excision sites will be randomly assigned to use the FS2 restorative wound care product on one excision site and a vehicle formulation of the product on the other. At the discretion of the Principal Investigator, a sutured wound may be bisected for intra-wound comparison of treatments. In all cases, after application of either vehicle or FS2, a layer of petrolatum will be applied to cover the wound site as a standard of care.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female
2. Adult, Senior (>18 years of age)
3. Healthy or medically stable
4. Requiring surgical removal (excision) of two (2) anatomically significantly similar areas and/or an excision of 3 - 10 cm in length suitable for intra-wound treatment comparison
5. Willing and able to follow study requirements

Exclusion Criteria:

1. Subjects who are medically unstable
2. Subjects who are expected to be medically unstable for the duration of the study period and an additional 1-month thereafter
3. Pregnant subjects, or those attempting to become pregnant
4. Subjects with known immunosuppression or immunosuppressive illness
5. Subjects with uncontrolled diabetes or autoimmune disorders
6. Subjects with known sensitivity to ingredients in the test-treatment products
7. Any other diagnosis, condition, physical or geographical limitation that may render, or increases the likelihood of rendering, the Subject unable to complete the entire study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-11-05 (Actual); Primary Completion 2020-09-29 (Actual); Study Completion 2020-09-29 (Actual)

PRIMARY OUTCOMES:
Vancouver Scar Scale (VSS) | 180 Days
  Investigator assessment of target scar or keloid using the Vancouver Scar Scale (VSS). Scale parameters include: Pigmentation (0-2), Vascularity (0-3), Pliability (0-5), and Height (0-3). Scale measurements include: minimum score of 0 = normal to a maximum score of 2, 3 or 5 depending on the parameter measured.
Patient and Observer Scar Assessment Scale (POSAS) | 180 Days
  Investigator assessment of target scar or keloid using the Patient and Observer Scar Assessment Scale (POSAS). Scale parameters include: Vascularity, Pigmentation, Thickness, Relief, Pliability, and Surface Area. Scale measurements include: minimum score of 1 = normal skin to a maximum score of 10 = worst scar imaginable.

CONTACTS AND LOCATIONS:
Overall Officials: Mark S Nestor, M.D., Ph.D., Principal Investigator — The Center for Clinical and Cosmetic Research
Locations (1):
- The Center for Clinical and Cosmetic Research, Aventura, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: BirchBioMed Inc. — http://www.birchbiomed.com